CLINICAL TRIAL: NCT06369454
Title: A PHASE 1, RANDOMIZED, OPEN-LABEL, 2-SEQUENCE, 3-PERIOD STUDY TO CHARACTERIZE THE GASTROINTESTINAL TRANSIT OF A MODIFIED-RELEASE CAPSULE FORMULATION UNDER FASTED AND FED CONDITIONS BY SINGLE LABEL GAMMA SCINTIGRAPHY IN HEALTHY MALE ADULT PARTICIPANTS
Brief Title: A Study to Learn About How Different Forms of the Study Medicine Called Ritlecitinib Pass the Intestines of Healthy Male Adults When Taken With or Without Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B7981090
Record Dates: First submitted 2024-04-11; First posted 2024-04-17 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics,; Scintigraphy,; Adults
MeSH Terms: interventions — PF-06651600

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence 1 (Experimental): Ritlecitinib 100 mg solution (fasted, Period 1), followed by ritlecitinib 100 mg MR capsule with 153Sm2O3 (fasted, Period 2), and followed by ritlecitinib 100 mg MR capsule with 153Sm2O3 (fed, Period 3).
  Interventions: Drug: Ritlecitinib
- Treatment Sequence 2 (Experimental): Ritlecitinib 100 mg solution (fasted, Period 1), followed by ritlecitinib 100 mg MR capsule with 153Sm2O3 (fed, Period 2), and followed by ritlecitinib 100 mg MR capsule with 153Sm2O3 (fasted, Period 3).
  Interventions: Drug: Ritlecitinib

INTERVENTIONS:
Drug: Ritlecitinib — Ritlecitinib 100 milligrams (mg) will be provided as either solution or capsule formulation (2 capsules of 50 mg) with 153Sm2O3
  Other Names: PF-06651600

SUMMARY:
The purpose of this study is to learn about how different forms of the study medicine called ritlecitinib pass the intestines of healthy male adults when taken with or without food.

This study is seeking healthy participants who have:

* Aged 18 years or older;
* male who are healthy as determined by medical assessment;
* BMI of 16-32 kg/m2, and a total body weight >45 kg (99 lb).

All participants in this study will receive a ritlecitinib oral dose in two different forms (solution without food, capsule with or without food).

The study will take up to 3 months, including the screening period and follow-up phone call. Participants will have to stay at the study clinic for at least 11 days. There will be 3 periods in total, and a washout period of at least 3 days between dosings in Period 1 and Period 2, and at least 7 days between dosings in Period 2 and Period 3 for this study. On day 1 of each period, participants will take one form of Riltecitinib without food for the first two periods and with food for the last period. Participants will have blood samples taken both before and after taking ritlecitinib. A follow-up phone call will be made at 28 to 35 days after the last study period.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants aged 18 years or older (or the minimum age of consent in accordance with local regulations) at screening who are overtly healthy as determined by medical evaluation including medical history, physical examination, and laboratory tests.
2. BMI of 16-32 kg/m2, and a total body weight >45 kg (99 lb).
3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
4. Capable of giving signed informed consent

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Participants with the acute or chronic infections or infection history
3. History of febrile illness within 5 days prior to the first dose of study intervention.
4. History of any lymphoproliferative disorder such as EBV related lymphoproliferative disorder, history of lymphoma, history of leukemia, or signs or symptoms suggestive of current lymphatic or lymphoid disease.
5. Known present or a history of malignancy other than a successfully treated or excised nonmetastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.
6. History of active or latent Mycobacterium TBA: participant who is currently being treated for active or latent Mycobacterium TB infection or has a history of Mycobacterium TB must be excluded from the study.
7. Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
8. Recent history of abnormal bowel movements, such as diarrhea, loose stools, or constipation, within 1 week prior to first dose.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2024-05-03 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Site of capsule disintegration and MR microsphere dispersion | up to 48 hours post dose or as long as radioactivity is present in the GI tract (if it is shorter than 48 hours)
  The time and gastrointestinal location where the HPMC capsule(s) disintegrate and disperse the drug formulation.
Gastric emptying time | up to 48 hours post dose or as long as radioactivity is present in the GI tract (if it is shorter than 48 hours)
  Gastric emptying metrics may include a) time of 1st GE; b) time(s) for GE 10%, 25%, 50%, 75%, 90% and complete gastric emptying time GE100%.
Small intestine residence/transit time | up to 48 hours post dose or as long as radioactivity is present in the GI tract (if it is shorter than 48 hours)
  Small Intestine transit metrics may include time for 10%, 25%, 50%, 75%, 90% and 100% of the formulation to transit through the small intestine.
Colon arrival time | up to 48 hours post dose or as long as radioactivity is present in the GI tract (if it is shorter than 48 hours)
  Arrival time at the colon (ATC) metrics may include a) time(s) for ATC 10%, 25%, 50%, 75%, 90% and 100%.
Colon (ascending, transverse, descending) residence/transit time | up to 48 hours post dose or as long as radioactivity is present in the GI tract (if it is shorter than 48 hours)
  The residence time of the formulation in the three primary regions of the large intestine to include the ascending, transverse and descending colon.
Total transit time | up to 48 hours post dose or as long as radioactivity is present in the GI tract (if it is shorter than 48 hours)
  Residence time of the formulation in the gastrointestinal tract.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | Solution: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post-dose. Capsules: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose.
  Maximum plasma concentration (Cmax)
Area under the plasma concentration-time profile from time zero extrapolated to infinite time (AUCinf) | Solution: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post-dose. Capsules: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose.
  Area under the plasma concentration-time profile from time zero extrapolated to infinite time (AUCinf) will be calculated if data permit.
Area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration (AUClast) | Solution: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post-dose. Capsules: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose.
  Area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration (AUClast)
Time for Cmax (Tmax) | Solution: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post-dose. Capsules: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose.
  Time for Cmax (Tmax)
Terminal half-life (t1/2) | Solution: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post-dose. Capsules: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose.
  Terminal half-life (t1/2) will be calculated if data permit.
Frequency of adverse events | Baseline up to Day 35
  To evaluate safety and tolerability of ritlecitinib following single oral administration as solution and MR capsule formulations in healthy male adult participants.
Frequency of abnormal clinical laboratory tests | Baseline up to Day 11
  To evaluate safety and tolerability of ritlecitinib following single oral administration as solution and MR capsule formulations in healthy male adult participants.
Frequency of abnormal vital signs | Baseline up to Day 11
  To evaluate safety and tolerability of ritlecitinib following single oral administration as solution and MR capsule formulations in healthy male adult participants.
Frequency of abnormal 12-lead ECG | Baseline up to Day 11
  To evaluate safety and tolerability of ritlecitinib following single oral administration as solution and MR capsule formulations in healthy male adult participants.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Scintipharma - Lexington - Maywick View Lane, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981090